CLINICAL TRIAL: NCT05439837
Title: Paracoracoid Subscapularis Plane Block Versus Infraclavicular and Subomohoid Block for Shoulder Surgery
Brief Title: Paracoracoid Subscapularis Plane Block Versus Iso Block for Shoulder Surgery for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Amr hamdy Mahmoud, Assistant lecturer of anesthesia and intensive care, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D 229
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infraclavicular and subomohoid block (Active Comparator)
  Interventions: Procedure: Infraclavicular and subomohoid block
- Paracoracoid subscapularis plane block (Active Comparator)
  Interventions: Procedure: Paracoracoid subscapularis plane block

INTERVENTIONS:
Procedure: Infraclavicular and subomohoid block — Its blockade of subscapular nerve in the subscapular fossa and axillary nerve as it curves around humeral And blocking of brachial plexuses cord and supra scapular nerve And blocking of the brachial plexuses cord and supra scapular nerve
  Arms: Infraclavicular and subomohoid block
Procedure: Paracoracoid subscapularis plane block — Blocking of suprascapular nerve in supra scapular fossa and axillary nerve as it curves the humeral head
  Arms: Paracoracoid subscapularis plane block

SUMMARY:
Shoulder surgery is the second orthopedic operation cause post operative pain Interscalene block is the standard block for shoulder surgery but it cause phrenic nerve block and diaphragmatic hemipareses Iso block is the block used to block the brachial plexuses cord and suprascapular nerve And paracoracoid subscapularis block supra scapular nerve in supra scapular fosa and axillary nerve as it curves around humeral head

DETAILED DESCRIPTION:
Two groups Group S for paracoracoid subscapularis block Group I for iso block Twenty patients for para coracoid subscapularis block with ultra sonography 50 mm 22G needle inserted anterior to the fascia and 15ml o.5% bupivicaine injected another twenty patients for iso block a linear probe of ultrasound is placed in the infraclavicular region to identify the cords the needle is inserted 2-3cm superior to the clavicle and advanced in.plane posterior to the clavicle toward the cods and 25ml local anaesthesia is injected

ELIGIBILITY:
Inclusion Criteria:

* male or female patient >20year for shoulder surgery American Society of anaesthesiologist physical state 1 to2

Exclusion Criteria:

* refusal of patient Systemic infection Local infection Neurological or respiratory disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment by VAS score | At 48 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Shawky, MD, Principal Investigator — Fayoum university hodpital; Joseph M Botros, MD, Principal Investigator — Eygpt fayoum university; Maged L Bolus, MD, Principal Investigator — Fayoum universty hospital
Locations (1):
- Fayoum University hospital, Al Fayyum, Fayoum, Madīnat Al Fayyūm, Faiyum Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garrett WE Jr, Swiontkowski MF, Weinstein JN, Callaghan J, Rosier RN, Berry DJ, Harrast J, Derosa GP. American Board of Orthopaedic Surgery Practice of the Orthopaedic Surgeon: Part-II, certification examination case mix. J Bone Joint Surg Am. 2006 Mar;88(3):660-7. doi: 10.2106/JBJS.E.01208. No abstract available. PMID 16510834